CLINICAL TRIAL: NCT04815473
Title: AndraValvulotome Post-Market Study
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: The number of evaluated valves were achieved.
Sponsor: Andramed GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VSP-001
Record Dates: First submitted 2021-03-19; First posted 2021-03-25 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients treated with AndraValvulotome (Other)
  Interventions: Procedure: Valvulotomy

INTERVENTIONS:
Procedure: Valvulotomy — Valvulotomy of the venous valves

SUMMARY:
The AndraValvulotome Post-Market Study is a prospective, open-label, multi-center study to evaluate the efficacy and safety of the AndraValvulotome. A maximum of 70 patients will be enrolled with peripheral artery disease (PAD) in up to 10 sites. Study participants will be primarily observed during the bypass procedure. In addition, the patients will be re-evaluated at the follow-up visit which will be scheduled 30 +/- 7 days after beginning of the study participation.

The objective of this study is to analyze the efficacy and safety of the valvulotomy of the venous valves with the CE marked AndraValvulotome during the bypass procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with peripheral arterial disease who are planned to undergo a bypass surgery with autologous vena saphena magna and using a valvulotome.
* Patient has to be consented and a informed consent form needs to be signed.
* Patient is able to and willing to participate in the 30 days follow-up.
* Vein diameter is at least 2mm (4F system) and 3mm (5F system).
* Vein diameter does not exceed 8mm (OTW-version) or 6mm (TIP-version)
* Bypass needs to be a continuous vena saphena magna with a length of at least 20cm.
* Rutherford category III - VI

Exclusion Criteria:

* Patients who have not completed 18 years of age
* Patients who are pregnant or assuming to be pregnant, and breast feeding.
* Patients who cannot participate due to medical or physical condition based on the decision of the physician.
* Life expectancy less than 1 year
* Known allergies to materials of the tip, cutting basket, outer catheter, kink protection and braid.
* Rutherford category 0-2
* Using varicose vein
* Exclusion criteria based on IFU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Absence of device related serious adverse events (SAE) | until 30 +/- 7 days follow-up visit
Rate of not sufficiently incised venous valves | Until approximately 10 days after procedure or discharge
Pulsatile blood flow | during procedure

SECONDARY OUTCOMES:
Quantity of device related bleeding | until 30 +/- 7 days follow-up visit
  A device related bleeding could occur due to the application of the device. Bleeding is defined as a decrease of a value of 2 hemoglobin points.
Severity of device related bleeding | until 30 +/- 7 days follow-up visit
  A device related bleeding could occur due to the application of the device. Bleeding is defined as a decrease of a value of 2 hemoglobin points.
Quantity of device related AE and SAE | until 30 +/- 7 days follow-up visit
Severity of device related AE and SAE | until 30 +/- 7 days follow-up visit
Quantity of passages of valvulotomy | during procedure
Primary patency rate | until 30 +/- 7 days follow-up visit
Primary technical success | Until approximately 10 days after procedure or discharge
  technical success is defined as clinical efficacy after valvulotomy without the presence of device related AE and SAE

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Hyhlik-Dürr, MD, Principal Investigator — University Clinic Augsburg
Locations (4):
- Germany (4):
  - University Clinic Augsburg, Augsburg
  - Evangelisches Krankenhaus Hubertus, Berlin
  - St. Bernward Krankenhaus, Hildesheim
  - University Clinic Leipzig, Leipzig